CLINICAL TRIAL: NCT03698110
Title: Programa Padres y Madres Unidos Educando en Estilos de Vida Saludables
Brief Title: Programa PUEDES Infancia
Acronym: PUEDES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Navarra (Other)
Responsible Party: Principal Investigator, Cayetana Ruiz Zaldibar, PhD in Nursing Student, University of Navarra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017.025
Record Dates: First submitted 2017-11-17; First posted 2018-10-05 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Parenting; Self Efficacy; Life Style

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participated in one introductory session, in the four sessions of PUEDES program during four weeks and in a closing session.
  Interventions: Behavioral: Intervention Group
- Control Group (No Intervention): Participated in one introductory session and in a closing session.

INTERVENTIONS:
Behavioral: Intervention Group — PUEDES program included eight hours in groups and activities to practice at home.
  Other Names: PUEDES program group
  Arms: Intervention Group

SUMMARY:
The purpose of this study was to evaluate whether an intervention directed at promoting parental self-efficacy and skills, based on a positive parenting framework, improves parental competences and healthy practices in families with children aged 2 to 5 years old.

DETAILED DESCRIPTION:
This study has designed implemented and evaluated an intervention to promote parental competence and healthy practices in families with children aged 2 to 5 years old, addressing parental self-efficacy an skills. This research followed the first three stages of the Medical Research Council framework for complex interventions: the theoretical, modeling and exploratory trial phases. A randomized control trial with parents of children better 2 to 5 years old was conducted. The program consisted of two hour long four sessions. Parents were grouped in small groups (7-8 participants) and guided by a facilitator whose role was to provide a participative and trusting atmosphere to share opinions and experience in healthy lifestyles and parenting. Data collection was performed at three time points (pre-intervention, post-intervention and follow-up) to asses the preliminary efficacy, acceptability and feasibility of the program.

ELIGIBILITY:
Inclusion Criteria:

* Be father or mother of at list one child between 2 to 5 years old
* Be over 18 years old
* Sign the informed consent

Exclusion Criteria:

* Fathers or mothers that could have special necessities that could prevent the course of the sessions
* Participants the could understand or speak spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-11-17 (Actual)

PRIMARY OUTCOMES:
Change from baseline Parental Self-efficacy at post-intervention and three months. Tool to Measure Parental Self-efficacy (TOPSE) is a questionnaire developed to measure parental self-efficacy. | baseline (before starting the program), post-intervention (5 weeks) and follow-up (3 months after the end of the program)
  Parenting self-efficacy (PSE) describes a parent's belief in their ability to perform the parenting role successfully. Tool to Measure Parental Self-efficacy (TOPSE) is specifically useful for the evaluation of parenting programs. TOPSE has 8 subscales about emotion and affection, play and enjoyment, empathy and understanding, control, discipline and boundaries, external pressures on parenting, acceptance of oneself and learning and knowledge.Regarding the validity and reliability of the scale varies between 0.80 and 0.89 per item, and of 0.94 as a whole (Kendall and Bloomfield, 2005).
Change from baseline Parenting styles at post-intervention and three months. Parenting styles scale is a validated tool to measure the different types of parenting styles (democratic, authoritative, permissive or negligent). | baseline (before starting the program), post-intervention (5 weeks) and follow-up (3 months after the end of the program)
  Parenting styles are the differences strategies that parents use in their child rearing. Parenting style scale called Escala de Evaluación de Estilos Educativos (4E), measures the different types of parenting styles (democratic, authoritative, permissive or negligent).It evaluates, through 20 items on a Likert scale the posture of parents in the traditional dimensions of educational styles: affection and communication, demands and control.The reliability coefficient of Cronbach's alpha of the scale is 0.73 (Sánchez-Sandoval, León and Román, 2012).
Change from baseline Parenting Practice in health promotion at post-intervention and three months. Meals in our household is a parent-report questionnaire that measures six domains related to the families' mealtimes. | baseline (before starting the program), post-intervention (5 weeks) and follow-up (3 months after the end of the program)
  They are difference practices that parents practice in there daily life that could promote healthy habits in their families.Questionnaire Meals in our household will be used to assess structure of family meals, problematic child mealtime behaviours, use of food as reward, parental concern about child diet, spousal stress related to child's mealtime behaviour, influence of child's food preferences on what other family members eat. The reliability coefficient of Cronbach's alpha is 0.77 (Anderson et al. 2012).
Change from baseline Parenting Practice in health promotion at post-intervention and three months. Comprehensive Feeding Practice is a questionnaire focused on parents practice related to meals. | baseline (before starting the program), post-intervention (5 weeks) and follow-up (3 months after the end of the program)
  Comprehensive Feeding Practice Questionnaire is reported by parents and assess the children involvement in meal planning and preparation and parental role model focused on if parents actively demonstrate healthy eating for the child.

SECONDARY OUTCOMES:
Parental satisfaction with the program. Questionnaire developed by researchers. | Post-intervention (5 weeks).
  Parents from the intervention group will be asked about their parental satisfaction with the program. Their opinion about its need, and whether they will be able to recommend it to friends or family, using a Likert scale of 0 to 10 developed by researchers, where 0 is nothing and 10 is completely, also were questions of this questionnaire.
Positive parenting program evaluation. The Evaluation system of positive parenting programs is a scale developed to assess positive parenting programs. | Post-intervention (5 weeks).
  The Evaluation system of positive parenting programs was designed to evaluate the interventions in positive parenting in Spain (Manzano et al., 2012). It is a tool that professional could use in the implementation, methodology and content of the program. The system has 17 indicators that refer to different aspects of intervention programs such as general assessment, objectives, materials, evaluation or ethical aspects. The results will be collected in a table that will show the scores of all the indicators, the total score of each thematic block and the final score obtained in the instrument. In this way it will be observed what parts of the program have more power and which should be improved.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kendall S, Bloomfield L. Developing and validating a tool to measure parenting self-efficacy. J Adv Nurs. 2005 Jul;51(2):174-81. doi: 10.1111/j.1365-2648.2005.03479.x. PMID 15963189
- [Background] Sánchez-Sandoval Y, León E, Román M. Adaptación familiar de niños y niñas adoptados internacionalmente. Anales de psicología 28(2): 558-566, 2012
- [Background] Anderson SE, Must A, Curtin C, Bandini LG. Meals in Our Household: reliability and initial validation of a questionnaire to assess child mealtime behaviors and family mealtime environments. J Acad Nutr Diet. 2012 Feb;112(2):276-84. doi: 10.1016/j.jada.2011.08.035. PMID 22741169
- [Background] Musher-Eizenman D, Holub S. Comprehensive Feeding Practices Questionnaire: validation of a new measure of parental feeding practices. J Pediatr Psychol. 2007 Sep;32(8):960-72. doi: 10.1093/jpepsy/jsm037. Epub 2007 May 28. PMID 17535817